CLINICAL TRIAL: NCT03907501
Title: The Effects of Organic Triphala and VSL#3 Probiotic Supplementation on Stool Microbiome Profiles and Inflammation in Healthy Elderly Subjects
Brief Title: Effects of Triphala and VSL#3 Probiotic Supplementation on Stool Microbiome Profiles and Inflammation
Acronym: TRIPH2017
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 related personnel, reagent and budget related impacts
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christine T. Peterson, Assistant Project Scientist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TRIPH2017
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Human Microbiome
Keywords: Gastrointestinal System; Inflammatory Biomarkers; Psychological Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Synbiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: Interested and eligible participants will be randomly assigned to either an 8-week synbiotic group, herb alone, or placebo control with a goal to obtain 60 patients who complete the study (20 in each group) after an estimated 20% attrition. Placebo control subjects will be given the option of having the 8-weeks of herbal synbiotic for directed personal use upon conclusion of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study will employ double-blind masking and only the project manager will be aware if the participant is assigned to take the synbiotic, triphala alone, or placebo. At the end of the 8 weeks, participants will be made aware of their randomly assigned supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synbiotic (Experimental): Two grams of organic Triphala powder (Banyan Botanicals, Inc.) with 1 capsule VSL#3® (VSL Pharmaceuticals, Inc.) probiotic taken with a few ounces of room temperature water in the morning and at bedtime for 8 weeks. Subjects will be provided both written and verbal instructions and given a kit containing encapsulated Organic Triphala powder (Banyan Botanicals, Inc.) and VSL#3® (VSL Pharmaceuticals, Inc.) capsules.
  Interventions: Dietary Supplement: Synbiotic
- Probiotic (Active Comparator): Subjects will be provided both written and verbal instructions and given a kit containing encapsulated Organic Triphala powder (Banyan Botanicals, Inc.). Subjects will take 2 grams of organic Triphala powder with a few ounces of room temperature water in the morning and at bedtime.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Subjects will be provided both written and verbal instructions and given a kit containing placebo capsules. Subjects will be instructed to take 2 (inert) capsules with room temperature water in the morning and at bedtime.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — an herbal prebiotic plus probiotic
  Arms: Synbiotic
Dietary Supplement: Probiotic — Triphala alone
  Arms: Probiotic
Dietary Supplement: Placebo — Inert capsule
  Arms: Placebo

SUMMARY:
Normal aging can lead to loss of gut microbial biodiversity which is linked to inflammaging and immunosenescence or the loss of immunocompetence. Probiotics, such as VSL#3®, and certain herbal supplements such as Triphala are associated with restoration of gut community architecture, increased gut barrier function and decreased inflammation. The present project will examine the potential benefits of a synbiotic (which denotes a prebiotic plus probiotic, and in this study, is an herbal prebiotic plus probiotic) intervention (8 weeks of supplementation) on gut microbiome profiles assessed via stool, inflammatory blood markers, and questionnaires about gastrointestinal health and mood. In this exploratory study, the investigators will examine psychological and physical functioning at baseline and after 8 weeks of supplementation with synbiotic, Triphala alone, or placebo.

DETAILED DESCRIPTION:
Primary Aim: In healthy, cognitively intact elderly subjects, determine the effects of an 8-week synbiotic supplement intervention on the stool microbiome (pre- and post-intervention) as compared to Triphala alone and placebo.

Secondary Aim: In healthy elderly subjects, examine the effects of an 8-week synbiotic supplementation intervention on inflammatory blood markers compared to herb alone or placebo.

Exploratory Aim 1: In healthy elderly subjects, examine the effects of an 8-week synbiotic intervention on gastrointestinal and psychological health via questionnaires compared to herb alone or placebo.

ELIGIBILITY:
Inclusion criteria:

1. Cognitively intact;
2. Able to give informed consent in English;
3. Medical clearance by their doctor;
4. > 60 years of age.

Exclusion criteria:

1. Alzheimer's Disease or other neurodegenerative disease such as Parkinson's Disease;
2. Current use or use in the past 3 months of antimicrobial or steroidal drugs;
3. Medical conditions affecting immune status (e.g., rheumatoid arthritis, heart failure, hepatitis C, HIV);
4. Individuals diagnosed with Diabetes Mellitus
5. International travel in past 3 months.
6. Previous known side effect or negative reaction to VSL#3 or Triphala

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine T Peterson, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates 07/01/2019 - 11/01/2019. The location is UCSD School of Medicine Building 4 via IRB approved phone script. 34 subjects were approved for enrollment for our first wave of intervention/subjects and 18 began the study before the study was closed.
Pre-assignment Details: 18 subjects began the intervention (2 dropped out) before the study was closed. Few subjects were able to begin the intervention compared to what was planned before the study was closed due to multiple pandemic related impacts. As the budget was impacted, no data was generated. No data is reported as the samples will not be processed and no data was generated.
Groups:
- Synbiotic: Synbiotic Group. Subjects will be provided both written and verbal instructions and given a kit containing encapsulated Organic Triphala powder (Banyan Botanicals, Inc.) and VSL#3® (VSL Pharmaceuticals, Inc.) capsules. Subjects will take 2 grams of encapsulated organic Triphala powder and 1 capsule of VSL#3 with room temperature water in the morning and at bedtime.
  Synbiotic: an herbal prebiotic plus probiotic
- Triphala: Triphala Group. Subjects will be provided both written and verbal instructions and given a kit containing Triphala capsules (Banyan Botanicals). Subjects will take 4 capsules (2g) of Triphala with room temperature water in the morning and at bedtime.
  Triphala: encapsulated
- Placebo: Subjects will be provided both written and verbal instructions and given a kit containing encapsulated placebo powder (made by VSL#3 manufacterer). Subjects will take 2 grams of organic placebo powder with a few ounces of room temperature water in the morning and at bedtime.
  Placebo: Inert capsule
Period: Overall Study
Arm/Group | Synbiotic | Triphala | Placebo
Started | 7 | 6 | 5
Completed | 6 | 5 | 5
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: As only a few subjects took the intervention before the study was closed due to COVID-19, no data was generated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Synbiotic | Triphala | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 5 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 2
  >=65 years | 6 | 5 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (5.0) | 74.5 (8.4) | 73.6 (6.6) | 72.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 4 | 3 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Measures of Gut Microbiome Health
Description: 16S rDNA sequencing of stool sample
Time Frame: 8 weeks
Population: Study closed due to COVID-19. No data was generated. No data was analyzed.
Groups:
- Triphala: Subjects will be provided both written and verbal instructions and given a kit containing encapsulated Organic Triphala powder (Banyan Botanicals, Inc.). Subjects will take 2 grams of organic Triphala powder with a few ounces of room temperature water in the morning and at bedtime.
  Probiotic: Triphala alone
Arm/Group | Synbiotic | Triphala | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Inflammatory Biomarkers
Description: Measure concentrations of 30 cytokines in blood samples with standard ELISA panel
Time Frame: 8 weeks
Population: No data was generated or analyzed. Study closed due to COVID-19 impacts.
Arm/Group | Synbiotic | Triphala | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months.
Description: Adverse event collection was obtained by the UCSD study coordinator and clinical attendants.
Groups:
- Probiotic: Probiotic Group. Subjects will be provided both written and verbal instructions and given a kit containing VSL#3® (VSL Pharmaceuticals, Inc.) capsules. Subjects will take 1 capsule of VSL#3 with room temperature water in the morning and at bedtime.
  Probiotic: capsule
Arm/Group | Synbiotic | Probiotic | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
Study Closed early due to COVID-19 related impacts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03907501/Prot_SAP_000.pdf